CLINICAL TRIAL: NCT07262268
Title: A Phase 1b, Double-Blind, Crossover Study of BHV-7000 in Patients With Inherited Erythromelalgia (IEM) With NaV1.7 Gain of Function Mutations
Brief Title: A Phase 1b Study of BHV-7000 in Participants With Inherited Erythromelalgia
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV7000-119
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Familial Erythromelalgia
Keywords: Erythomelalgia; IEM; Primary Erythomelalgia; SCN9A; NaV1.7; Channelopathy; Red Neuralgia; Neuropathic Pain; Inherited Erythomelalgia
MeSH Terms: conditions — Erythromelalgia; Generalized Epilepsy With Febrile Seizures Plus, 7; Channelopathies; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV-7000 (Experimental)
  Interventions: Drug: BHV-7000
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-7000 — Participants will take blinded investigational product (IP) orally once daily
  Other Names: opakalim
  Arms: BHV-7000
Drug: Placebo — Matching placebo taken orally once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the potential benefits of BHV-7000 in reducing chronic pain in participants with IEM with a previously demonstrated gain of function mutation in the SCN9A gene.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult men and women between 18 to 75 years of age, inclusive, at time of consent with a diagnosis of inherited erythromelalgia with a previously characterized gain of function NaV1.7 mutation resulting in chronic pain.
2. Absence of concomitant mutation resulting in Kv7.2/7.3 gain of function.
3. Ability and willingness to adhere to the study procedures and complete accurate pain diaries
4. Stable background analgesic regimen for at least 30 days before screening and willingness to maintain the same analgesic regimen during the study period.

Key Exclusion Criteria:

1. Any clinically significant laboratory abnormalities or clinically significant abnormalities on screening physical examination, vital signs, or ECG that, in the judgment of the principal investigator, indicates a medical problem that would preclude study participation.
2. Any medical condition, based on the judgement of the Investigator, that would confound the ability to adequately assess safety and efficacy outcome measures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean of the daily average maximum pain intensity scores collected every 2 hours. | The last 3 weeks of each 4-week crossover treatment period
  Participants will be asked to record peak (worst) pain experienced in the previous 2 hours using an 11-point Likert scale (0-10) where 0=no pain and 10=worst possible pain

SECONDARY OUTCOMES:
The average weekly frequency of pain attacks on treatment vs. placebo | The last 3 weeks of each 4-week crossover treatment period
  Participants will be asked to record occurrence of pain attacks
The average duration of pain attacks on treatment vs. placebo | The last 3 weeks of each 4-week crossover treatment period
  Participants will be asked to record the duration of their pain attacks
The average peak severity of pain attacks on treatment vs. placebo | The last 3 weeks of each 4-week crossover treatment period
  Participants will be asked to record the maximum severity of their pain attacks using an 11-point Likert scale (0-10) where 0=no pain and 10=worst possible pain.
Safety and tolerability by reporting the frequency of unique participants with SAEs, severe AEs, AEs leading to discontinuation, deaths, and Grade 3-4 (CTCAE/DAIDS) laboratory abnormalities. | Up to 16 weeks
  Measured by assessing the number of unique participants who experience treatment-emergent serious adverse events, adverse events leading to discontinuation, or moderate and severe adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Site-001, New Haven, Connecticut, United States